CLINICAL TRIAL: NCT04617782
Title: A Phase 1, Open-Label, 3-Period, Randomized, Crossover Pharmacokinetic Study to Evaluate the Steady-State Pharmacokinetics of 5 mg and 10 mg Corplex™ Donepezil TDS Compared to 10 mg Oral Aricept® in Healthy Volunteers
Brief Title: Pharmacokinetic Study of 5 and 10 mg Corplex™ Donepezil TDS Compared to 10 mg Aricept® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CL-P-20003
Record Dates: First submitted 2020-11-01; First posted 2020-11-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Healthy Subjects
Keywords: Donepezil, Transdermal Delivery System
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: Phase 1, open-label, randomized, 3-period, 3-treatment, crossover PK study to evaluate the steady-state pharmacokinetics
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): 5 mg/day Donepezil Transdermal Delivery System (TDS) 1-week wear and applied weekly for 5 consecutive weeks
  Interventions: Combination Product: Donepezil TDS
- Treatment B (Experimental): 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks
  Interventions: Combination Product: Donepezil TDS
- Treatment C (Active Comparator): 10 mg/day Aricept® donepezil tablet administered QD for 5 consecutive weeks
  Interventions: Drug: Aricept

INTERVENTIONS:
Combination Product: Donepezil TDS — Transdermal Delivery System
  Arms: Treatment A; Treatment B
Drug: Aricept — Oral
  Arms: Treatment C

SUMMARY:
Phase 1, open-label, randomized, 3-period, 3-treatment, crossover pharmacokinetic study to evaluate the steady-state pharmacokinetics of 5 mg/day and 10 mg/day Corplex™ Donepezil TDS manufactured with the commercial process compared to 10 mg Aricept® in healthy volunteers.

DETAILED DESCRIPTION:
Screening Period:

Subjects will undergo a Screening Period up to 28 days prior to entering the Treatment Phase.

Treatment Phase consisting of 3 Treatment periods with 3 Treatments A, B, C.

Treatment Period 1: All Subjects will receive Treatment A; 5 mg/day Donepezil Transdermal Delivery System (TDS); 1-week wear and applied for 5 consecutive weeks.

Treatment Periods 2 and 3: Subjects will be randomized (by gender) to receive either sequences of Treatments B-C or Treatments C-B.

Treatment B: 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks Treatment C: 10 mg/day Aricept® donepezil tablet administered daily (QD) for 5 weeks.

Blood samples for pharmacokinetics and safety assessments will be collected during the Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females.
* Subject's Body Mass Index (BMI) must be between 18 and 32 kg/m2 (inclusive).
* Subject must be continuous non-smokers.
* Subject must have a Fitzpatrick skin type of I, II or III.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* After resting seated for at least 3 minutes, subjects should be excluded from the study with the following vital signs at Screening

  1. systolic blood pressure outside the range of 90-145 mmHg, or
  2. diastolic blood pressure outside the range of 50-90 mmHg, or
  3. resting heart rate outside the range of 40-100 beats per minute.
* Has an isolated ALT ≥1.5x the ULN or AST ≥1.5x the ULN at Screening; or both ALT and AST exceeding the ULN.
* Estimated creatinine clearance at screening <70 mL/min/1.73 m2.
* Prolonged corrected QT (Fridericia) on screening ECG (≥450 ms for both females and males).
* History or presence of excessive hairy skin on application sites as deemed by the Investigator to potentially interfere with patch adhesion or drug absorption.
* History or presence of significant skin damage, diffuse skin diseases-, scars, tattoos on the application sites or other skin disturbances as deemed by the Investigator to potentially interfere with drug absorption or skin tolerability assessments
* Use of donepezil hydrochloride or related drugs within 60 days prior to the first study drug administration.
* Has participated in another clinical trial within 30 days prior to Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bass, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

REFERENCES:
- [Derived] Tariot PN, Braeckman R, Oh C. Comparison of Steady-State Pharmacokinetics of Donepezil Transdermal Delivery System with Oral Donepezil. J Alzheimers Dis. 2022;90(1):161-172. doi: 10.3233/JAD-220530. PMID 36120781

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence ABC or ACB in Crossover Fashion: All subjects were assigned to receive all treatments, with a different sequence in treatment periods 2 and 3.
  Treatment A: 5 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout; Treatment B: 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout; Treatment C: 10 mg/day Aricept® donepezil tablet administered QD for 5 consecutive weeks, then 1 day washout;
Period: Treatment A - 5 mg TDS
Arm/Group | Treatment Sequence ABC or ACB in Crossover Fashion
Started (The disposition summary reported in the CSR does not list disposition by sequence of treatment, and instead lists disposition by the treatment received. The statistical group that analyzed the data was an external vendor that is no longer contracted and not available to re-analyze the participant flow by sequence. Since the Sponsor does not have internal statistical capabilities, the participant flow summary is presented by treatment received, and not by sequence of treatment.) | 60
Completed | 57
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — failure to follow site rules | 1
Period: Treatment B - 10 mg TDS
Arm/Group | Treatment Sequence ABC or ACB in Crossover Fashion
Started (The disposition summary reported in the CSR does not list disposition by sequence of treatment, and instead lists disposition by the treatment received. The statistical group that analyzed the data was an external vendor that is no longer contracted and not available to re-analyze the participant flow by sequence. Since the Sponsor does not have internal statistical capabilities, the participant flow summary is presented by treatment received, and not by sequence of treatment.) | 55
Completed | 53
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment C - 10 mg Oral
Arm/Group | Treatment Sequence ABC or ACB in Crossover Fashion
Started (The disposition summary reported in the CSR does not list disposition by sequence of treatment, and instead lists disposition by the treatment received. The statistical group that analyzed the data was an external vendor that is no longer contracted and not available to re-analyze the participant flow by sequence. Since the Sponsor does not have internal statistical capabilities, the participant flow summary is presented by treatment received, and not by sequence of treatment.) | 56
Completed | 53
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — failure to follow site rules | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were assigned to receive treatment sequence ABC or ACB in a crossover fashion.
  Treatment A: 5 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout; Treatment B: 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout; Treatment C: 10 mg/day Aricept® donepezil tablet administered QD for 5 consecutive weeks, then 1 day washout;
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black of African American | 3
  Race: Asian | 1
  Race: White | 56
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax)
Description: To evaluate steady-state donepezil plasma exposure (Cmax) following 5 weeks of treatment.
Time Frame: 35 days of each Treatment
Population: all subjects without major protocol deviations that could affect PK and who had at least one PK parameter derived
Measure: Mean (Standard Deviation); unit: Cmax ng/ml
Groups:
- Treatment A 5 mg TDS: Treatment A: 5 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout;
- Treatment B 10 mg TDS: Treatment B: 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout;
- Treatment C 10 mg Oral: Treatment C: 10 mg/day oral donepezil tablet administered QD for 5 consecutive weeks, then 1 day washout;
Arm/Group | Treatment A 5 mg TDS | Treatment B 10 mg TDS | Treatment C 10 mg Oral
Number analyzed (Participants) | 60 | 55 | 56
Cmax ng/ml | 29.9 (9.1) | 62.4 (19.9) | 70.5 (19.4)

2. Primary Outcome: Area Under the Curve (AUC)
Description: To evaluate steady-state donepezil plasma exposure (AUC) following 5 weeks of treatment
Time Frame: 35 days each Treatment
Population: all subjects without major protocol deviations that could affect PK and who had at least one PK parameter derived
Measure: Mean (Standard Deviation); unit: AUC h*ng/mL
Groups:
- Treatment A 5 mg TDS: Treatment A: 5 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout
- Treatment B 10 mg TDS: Treatment B: 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout
- Treatment C 10 mg Oral: Treatment C: 10 mg/day oral donepezil tablet administered QD for 5 consecutive weeks, then 1 day washout
Arm/Group | Treatment A 5 mg TDS | Treatment B 10 mg TDS | Treatment C 10 mg Oral
Number analyzed (Participants) | 60 | 55 | 56
AUC h*ng/mL | 4366.0 (1380.1) | 9099.0 (2972.1) | 8462.6 (2558.0)

ADVERSE EVENTS:
Time Frame: Collected from first dose of the study drug to last treatment day, 36 days per intervention for a total of 108 days
Groups:
- Treatment A - 5 mg TDS; Treatment B - 10 mg TDS; Treatment C - 10 mg Oral: Participants received treatment sequence ABC or ACB in a randomized, crossover fashion.
  Treatment A: 5 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout; Treatment B: 10 mg/day Donepezil TDS 1-week wear and applied weekly for 5 consecutive weeks, then 1 day washout; Treatment C: 10 mg/day oral donepezil tablet administered QD for 5 consecutive weeks, then 1 day washout;
Arm/Group | Treatment A - 5 mg TDS | Treatment B - 10 mg TDS | Treatment C - 10 mg Oral
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 32/60 | 30/55 | 32/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A - 5 mg TDS (N=60) | Treatment B - 10 mg TDS (N=55) | Treatment C - 10 mg Oral (N=56)
Constipation (Gastrointestinal disorders) | 9 | 3 | 10
Nausea (Gastrointestinal disorders) | 4 | 1 | 17
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 7
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3
Application Site Pruritis (General disorders) | 12 | 5 | 0
Application Site Dermatitis (General disorders) | 5 | 3 | 1
Fatigue (General disorders) | 2 | 1 | 5
Application Site Irritation (General disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 8 | 8 | 7
Dizziness (Nervous system disorders) | 3 | 2 | 11
Somnolence (Nervous system disorders) | 0 | 0 | 6
Insomnia (Psychiatric disorders) | 4 | 4 | 0
Nightmare (Psychiatric disorders) | 5 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT04617782/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04617782/SAP_001.pdf